CLINICAL TRIAL: NCT06495671
Title: Australasian Nanoparticle-mediated Magnetically Enhanced Diffusion for Ischemic Stroke (AusNanoMED)
Brief Title: Australasian Nanoparticle-mediated Magnetically Enhanced Diffusion for Ischemic Stroke
Acronym: AusNanoMED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Monash University (Other); Euphrates Vascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBC2402
Record Dates: First submitted 2024-06-26; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Stroke; Stroke
Keywords: thrombolysis; thrombolytic; endovascular thrombectomy; nanoparticle; magnetically enhanced diffusion; digital subtraction angiography
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: Bayesian optimal phase 2 trial
Masking Description: Primary outcome assessed by blinded imaging core laboratory. Day 90 modified Rankin scale assessed by central blinded clinician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Magnetically enhanced diffusion (Experimental): Intra-arterial iron nanoparticles (4 x 1mg doses delivered every 3 minutes) delivered via microcatheter proximal to site of arterial occlusion(s) with external rotating magnet, total procedure 30min.
  Interventions: Device: Magnetically enhanced diffusion

INTERVENTIONS:
Device: Magnetically enhanced diffusion — Iron nanoparticle (intra-arterial) + External magnet workstation
  Other Names: PULSE Nanomed System

SUMMARY:
Rapidly restoring blood flow to the brain in patients with stroke caused by a blocked blood vessel in the brain is the key to reducing disability. Current treatments often leave small blocked arteries that cannot be safely opened with mechanical clot removal devices. Furthermore, stagnant flow limits access of clot-dissolving medication to the clot. This trial tests iron nanoparticles (similar to iron infused to replace low body stores but injected directly into the brain artery upstream of the blockage) combined with an external rotating magnet that draws the nanoparticles towards the clot, overcoming stagnant blood flow. The aim is to bring fresh blood which contains naturally-occurring clot-dissolving substances, and any clot-dissolving medication that may be circulating, to the surface of the clot with the aim of restoring blood flow to the brain. The trial will recruit up to 30 patients. All will receive injection of nanoparticles via an angiogram (small tube inserted into a leg or arm artery and fed up into the brain artery under Xray control). The procedure takes 30min and the degree of success in opening the artery at the end of procedure is the primary outcome, combined with an absence of symptomatic brain bleeding at 24h.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with ischemic stroke within 24 hours of the time they were last known to be well
* Patient's age is ≥18 years
* Legal requirements for consent as per local legislative requirements are satisfied.
* Distal medium vessel intracranial arterial occlusion visible on CT-angiography, MR-angiography or catheter digital subtraction angiography (DSA) in the middle cerebral, anterior or posterior cerebral artery. The occlusion may be primary or secondary (ie following initial mechanical thrombectomy of a large vessel occlusion)

Exclusion Criteria:

* Intracranial hemorrhage (ICH) identified by CT or MRI
* Rapidly improving symptoms at the discretion of the investigator
* Pre-stroke mRS score of ≥ 3 (indicating functional dependence)
* Frank hypodensity in >1/3 of the affected arterial territory on non-contrast CT
* CT Perfusion ischemic core volume > 100 ml
* Known automated implantable cardiac defibrillator, pacemaker, cerebral aneurysm clip, cochlear implant, cranial neurostimulator or other device implant that is incompatible with the external magnetic field
* Known allergy or sensitivity to iron
* Known hemochromatosis, or known liver disease such as cirrhosis.
* Known aortic dissection
* Suspected septic embolization
* Contra indication to imaging with contrast agents
* Pregnant or lactating women
* Any terminal illness such that patient would not be expected to survive more than 6 months
* Current participation in another investigational drug or device treatment study
* Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with substantial reperfusion at final angiography (15 +/- 5min after final nanoparticle injection) without symptomatic intracranial hemorrhage on CT/MRI at 24h | 24 hours +/- 6 hours
  * Substantial reperfusion is defined as >50% reperfusion of the target occluded vessel territory at cerebral angiogram 15 (+/- 5) minutes after completion of the final nanoparticle injection. Target occluded vessel territory is defined based on the angiogram immediately prior to nanoparticle injection, as adjudicated by the core laboratory.
  * Symptomatic intracranial hemorrhage is defined according to the Heidelberg Classification as new intracranial hemorrhage detected by brain imaging within 24h associated with any of the items below in the absence of an alternative explanation for clinical deterioration:
    * ≥4 point increase in NIHSS at the time of diagnosis compared to the most recent NIHSS prior to worsening
    * ≥2 point increase in one NIHSS category
    * Leading to intubation/hemicraniectomy/external ventricular drain placement or other major medical/surgical intervention

OTHER OUTCOMES:
The proportion of participants with >90% reperfusion of the target occluded vessel territory at cerebral angiogram 15 (+/- 5) minutes after completion of the final nanoparticle injection | 15 minutes +/- 5 minutes after completion of the final nanoparticle injection
  - Near-complete reperfusion is defined as >90% reperfusion of the target occluded vessel territory at cerebral angiogram 15 (+/- 5) minutes after completion of the final nanoparticle injection. Target occluded vessel territory is defined based on the angiogram immediately prior to nanoparticle injection, as adjudicated by the core laboratory
Symptomatic intracranial hemorrhage | 24 hours +/- 6 hours
  - Symptomatic intracranial hemorrhage is defined according to the Heidelberg Classification as new intracranial hemorrhage detected by brain imaging within 24h associated with any of the items below in the absence of an alternative explanation for clinical deterioration:
  * ≥4 point increase in NIHSS at the time of diagnosis compared to the most recent NIHSS prior to worsening
  * ≥2 point increase in one NIHSS category
  * Leading to intubation/hemicraniectomy/external ventricular drain placement or other major medical/surgical intervention
Procedural arterial perforation | 24 hours +/- 6 hours
  Procedural arterial perforation that results in visible extravasation of contrast into the subarachnoid space
Death due to any cause | 90 days +/- 7 days
  Death due to any cause within 90 days
modified Rankin Scale (mRS) at 3 months | 90 days +/- 7 days
  Modified Rankin Scale ranges from 0 (no symptoms of stroke) to 6 (death), high scores indicate worse outcome. Outcome is descriptive and ordinal analysis compared to historical control (adjusted for baseline NIHSS and age).
modified Rankin Scale (mRS) 0-1 or no change from baseline at 3 months | 90 days +/- 7 days
  Modified Rankin Scale ranges from 0 (no symptoms of stroke) to 6 (death), high scores indicate worse outcome. Outcome is descriptive and compared to historical control (adjusted for baseline NIHSS and age).
modified Rankin Scale (mRS) 0-2 or no change from baseline at 3 months | 90 days +/- 7 days
  Modified Rankin Scale ranges from 0 (no symptoms of stroke) to 6 (death), high scores indicate worse outcome. Outcome is descriptive and compared to historical control (adjusted for baseline NIHSS and age).
Early neurological improvement | 3 days +/- 1 day or discharge if earlier
  8 point reduction in National Institutes of Health Stroke Scale (NIHSS) score or reaching 0-1 at 3 days. NIHSS ranges from 0-42 with higher scores representing more severe stroke. Outcome is descriptive and compared to historical control (adjusted for baseline NIHSS and age).
Reperfusion at 24 hours | 24 hours +/- 6 hours
  Resolution of perfusion lesion (<5mL region of brain with hypoperfusion defined as Tmax delay >6 sec) at 24 hours
Recanalization at 24 hours | 24 hours +/- 6 hours
  Resolution of arterial occlusion at 24 hours assessed using the arterial occlusive lesion (AOL) scale 3. AOL ranges from 0 (no recanalization) to 3 (complete recanalization).

CONTACTS AND LOCATIONS:
Overall Officials: Bruce CV Campbell, MBBS FRACP, Principal Investigator — University of Melbourne; Ronil V Chandra, MBBS FRANZCR, Principal Investigator — Monash University
Locations (7):
- Australia (7):
  - John Hunter Hospital, Newcastle, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - The Austin Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No